CLINICAL TRIAL: NCT01419873
Title: Pilot Study of a Model-based Approach to Blood Glucose Control in Very-low-birthweight Neonates
Brief Title: Study of a Model-based Approach to Blood Glucose Control in Very-low-birthweight Neonates
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Christchurch Women's Hospital (Other)
Responsible Party: Principal Investigator, Adrienne Lynn, Dr Adrienne Lynn, Christchurch Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URA/08/06/039
Record Dates: First submitted 2011-08-12; First posted 2011-08-18 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Hyperglycaemia
Keywords: Hyperglycaemia; Very low birthweight infants; Insulin
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Actrapid Human Insulin — Actrapid Insulin is a drug used in routine neonatal practice to treat hyperglycaemia. The intervention in this study was to base dosing on insulin by a computer based-model approach as opposed to sliding scales, fixed protocols or clinician intuition

SUMMARY:
Very low birthweight neonates commonly develop high blood sugar levels. There is an association between high blood sugar levels and poorer short term outcomes but it is not known whether the high sugar level itself actually causes the problems.

There are a range of ways to manage high sugar levels but there are no consensus guidelines to follow. One option is to manage the high sugar levels with an infusion of insulin. Studies looking at insulin infusions have often used fixed protocols to guide the amount of insulin to be given and are often complicated by hypoglycaemia.

This study investigated whether using a model-based approach to individualise insulin administration to neonates with high sugar levels would provide a safe and effective management option for controlling blood sugar levels and avoid the complication of low blood sugar levels.

ELIGIBILITY:
Inclusion Criteria:

* Birthweight <1500g
* Blood sugar >/= 10mmol/L
* Clinician decision to start an insulin infusion

Exclusion Criteria:

* Infants who were moribund and not expected to survive

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Hypoglycaemia whilst receiving insulin | Length of hospital stay in NICU which will be from birth to 5 months of age
  Hypoglycaemia whilst the patient is receiving insulin as per the model-based method will be documented. The patients may require insulin at any time in their admission to NICU from birth to a maximum of 5 months of age when they would no longer be admitted to NICU.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne M Lynn, FRACP, Principal Investigator — Canterbury District Helath Board
Locations (1):
- Christchurch Womens Hospital, Canterbury District Health Board, Christchurch, New Zealand

REFERENCES:
- [Derived] Le Compte AJ, Lynn AM, Lin J, Pretty CG, Shaw GM, Chase JG. Pilot study of a model-based approach to blood glucose control in very-low-birthweight neonates. BMC Pediatr. 2012 Aug 7;12:117. doi: 10.1186/1471-2431-12-117. PMID 22871230